CLINICAL TRIAL: NCT02021578
Title: Family Cognitive Behavioral Prevention of Depression in Youth and Parents
Brief Title: A Family Depression Prevention Program
Acronym: FDP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: San Diego State University (Other)
Responsible Party: Principal Investigator, Judith Garber, Professor, Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 8482529
Record Dates: First submitted 2013-12-19; First posted 2013-12-27 (Estimated); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Depression
Keywords: Depression; Mood disorder
MeSH Terms: conditions — Depression; Mood Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Interviewers who assess diagnostic outcomes are masked to participant condition.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Family Cognitive Behavioral Prevention (Experimental): A family cognitive behavioral program for parents and children. Parents learn parenting skills and cognitive behavioral techniques for managing depression. Children learn coping skills.
  Interventions: Behavioral: Family Cognitive Behavioral Prevention
- Written Information (Active Comparator): Families receive written materials about depression and the effects of parental depression on children.
  Interventions: Behavioral: Written information

INTERVENTIONS:
Behavioral: Family Cognitive Behavioral Prevention — Parent training and cognitive behavioral intervention with parents. Coping skills training with children.
  Other Names: Cognitive behavioral intervention; Coping skills training; Parent training
  Arms: Family Cognitive Behavioral Prevention
Behavioral: Written information — Reading materials about depression
  Other Names: Psychoeducation; Self-help
  Arms: Written Information

SUMMARY:
The primary aim is to prevent depression in youth and parents in a single, integrated family intervention.

Hypothesis 1a: Children in the Family Depression Prevention (FDP) program will have significantly lower levels of anxious/depressive symptoms and fewer onsets of depressive episodes as compared to children in the Written Information (WI) condition.

Hypothesis 1b: In parents, the amount of time in a depressive episode will be significantly lower for those in the FDP program as compared to those in the WI condition.

DETAILED DESCRIPTION:
Depression is a major public health problem affecting over 15 million U.S. adults annually and is especially prevalent in those of parenting age. Offspring of depressed parents are at increased risk of depression and therefore are a critical target for preventive interventions. The current study aims to reduce the rate of depression in parents and their children by adopting an innovative, family-based approach to simultaneously preventing depression in at-risk youth and in their affected parents. The rationale for this approach is based on (a) a conceptual model that integrates parenting processes, stress (particularly that which is associated with parental depression), and children's self-regulatory skills in the face of stress, (b) evidence that depression runs in families, (c) promising results from family- and child-focused depression prevention programs, (d) evidence that in adults, cognitive-behavioral therapy (CBT) reduces both depressive episodes and their recurrence, and (e) growing consensus among scientists, clinicians, and policymakers on the need for family-based models of healthcare. This 5- year, two-site randomized controlled trial will test a Family Depression Prevention (FDP) program for children (ages 9-15) and their parents with depressive disorders (past or current). This "dual prevention" approach is a novel synthesis of existing evidence-based intervention techniques drawn from child prevention and adult treatment models. Participating families (N=300) will be randomized to either FDP (10 weekly + 3 monthly sessions) or a written information comparison (WI) condition. All parents and children will be evaluated at pre- and post-intervention, and at 6-, 12-months from baseline.

ELIGIBILITY:
Inclusion Criteria:

* Parent with a current or history of a depressive disorder within child's life
* Children ages 9- to 15-years-old

Exclusion Criteria:

* Bipolar I (parent or child)
* Schizophrenia (parent or child)
* Current alcohol or drug abuse (parent or child)
* Conduct disorder; developmental disability (child)
* Current diagnosis of a depressive disorder (child)

Ages: 9 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 304 (Actual)
Dates: Start 2014-08-01 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
In children, the primary outcome is level of symptoms on the Youth Self-report form. | twelve months post baseline
  For child participants, we will assess change in their levels of symptoms on the Youth Self-report form at 12-month follow-up. T-scores range from 0 to 100; higher scores indicate more symptoms (i.e., worse outcome).

SECONDARY OUTCOMES:
In children, level of internalizing and externalizing symptoms on the Child Behavior Checklist completed by parent about the child | 12 months
  For child participants, we will assess change in their levels of symptoms on the Child Behavior checklist at 12-month follow-up.
Parents: Patient Health Questionnaire - 9 (PHQ-9) | 12 months
  Parent participants: The PHQ-9 measures 9 symptoms of depression on a 4-point scale. Scores can range from 0 to 36.
Children: depressive diagnoses | 12 months
  Children and parents are interviewed about the child's depressive symptoms with the Longitudinal Interval Follow-up Evaluation, which yields scores 1-6 for each week.

CONTACTS AND LOCATIONS:
Overall Officials: Judy Garber, PhD, Principal Investigator — Vanderbilt University; Bruce Compas, PhD, Principal Investigator — Vanderbilt University; Robin Weersing, PhD, Principal Investigator — San Diego State University
Locations (2):
- United States (2):
  - San Diego State University, San Diego, California
  - Vanderbilt University, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data reported in publications will be made available to researchers upon request.
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: Data will be available after publication of results.
Access Criteria: Written requests for specific data, hypotheses, and data analytic plan

REFERENCES:
- [Background] Kado-Walton M, Vreeland A, Henry L, Gruhn M, Compas B, Garber J, Weersing VR. Racial/ethnic differences in parenting behaviors among depressed parents. J Fam Psychol. 2023 Sep;37(6):763-773. doi: 10.1037/fam0001125. Epub 2023 Jun 26. PMID 37358525
- See also: Link to PMC10613481 — http://pubmed.ncbi.nlm.nih.gov/37358525/